CLINICAL TRIAL: NCT02878096
Title: An Open-Label, 2-Part Sequential Dose Study Designed to Assess the Absolute Bioavailability, Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-SK-1404 Administered to Healthy Male Subjects
Brief Title: Bioavailability of [14C]-SK-1404 ADME & IV Microtracer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QCL117764
Record Dates: First submitted 2016-08-05; First posted 2016-08-25 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Nocturia
Keywords: nocturnal polyuria
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [14C]-SK-1404 (Experimental)
  Interventions: Drug: [14C]-SK-1404

INTERVENTIONS:
Drug: [14C]-SK-1404 — In Part 1, each subject will receive a single PO dose of SK-1404 followed by an IV microtracer dose of [14C]-SK-1404.

SUMMARY:
The primary objectives of the study are:

* To determine the absolute bioavailability of SK-1404
* To assess the mass balance recovery after a single oral (PO) dose of carbon-14 (14C)-SK-1404
* To provide plasma, urine and faecal samples for metabolite profiling and structural identification

The secondary objectives of the study are:

* To determine the routes and rates of elimination of [14C]-SK-1404
* To identify the chemical structure of each metabolite with an exposure (AUC) of more than 10% of circulating total radioactivity
* To explore the intravenous (IV) pharmacokinetics (PK) of [14C]-SK-1404
* To further explore the PO PK of SK-1404
* To provide additional safety and tolerability information for SK-1404

DETAILED DESCRIPTION:
This is a single-centre, 2-part, open-label, non-randomised, sequential, single dose study in healthy male subjects. It is planned to enrol a single cohort of 6 healthy male subjects who will participate in Parts 1 and Part 2 of the study.

In Part 1, each subject will receive a single PO dose of SK-1404 followed by an IV microtracer dose of [14C]-SK-1404.

In Part 2, each subject will receive a single PO dose of [14C]-SK-1404.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 30 to 65 years of age
3. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)
7. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Males with pregnant partners
2. Participation in a clinical research study within the 3 months prior to IMP dose
3. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
4. Subjects who have previously been enrolled in this study
5. Subjects who have previously been dosed with SK-1404
6. History of any drug or alcohol abuse in the past 2 years
7. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine) in the past year
8. Current smokers and those who have smoked within the last 12 months; this includes cigarettes, e-cigarettes and nicotine replacement products. A breath carbon monoxide reading of greater than 10 ppm at screening or admission
9. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
10. Subjects who have been enrolled in an ADME study in the last 12 months
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
12. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
13. Aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase >1.5 × upper limit of normal confirmed by repeat testing
14. Serum sodium below the lower limit of normal

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) calculated with the AUC values of IV administration in Part 1 and PO administration in Part 2 | Predose to 96hr
Mass balance recovery of total radioactivity in urine, faeces and all excreta | Predose to 168hr
  Amount excreted (Ae), and Ae as a percentage of the administered dose (%Ae), cumulative recovery (Cum Ae) and cumulative recovery expressed as a percentage of the dose (Cum %Ae)
Number and structural identification of known and unknown metabolites of SK-1404 in the plasma, urine and faeces samples | Predose to 168hr

SECONDARY OUTCOMES:
Ae total radioactivity in plasma by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
%Ae total radioactivity in plasma by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
Cum Ae (total) for urine by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
Cum %Ae (total) for urine by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
Cum Ae (total) for faeces by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
Cum %Ae (total) for faeces by metabolite profiling and structural identification to estimate the routes and rates of elimination of [14C]-SK-1404 | Predose to 168hr
Number and structural identification of unknown metabolites of SK-1404 with an AUC of more than 10% of circulating total radioactivity | Predose to 168hr
The peak plasma concentration (Cmax) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The time from dosing at which Cmax was apparent (Tmax) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The elapsed time from dosing at which the analyte was first quantifiable in a concentration vs time profile (Tlag) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The area under the concentration-time curve from dosing to the last measurable concentration (AUC(0-last)) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The area under the concentration-time curve from dosing extrapolated to infinity (AUC(0-inf)) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The percentage of AUC(0-inf) extrapolated beyond the last measured time point (AUC%extrap) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The terminal elimination rate constant calculated from the slope of the apparent elimination phase (lambda-z) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent terminal elimination half-life (T1/2) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent total clearance (CL/F) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent volume of distribution (Vd) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent volume of distribution (Vss) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The mean residence time (MRT) of SK-1404F and its active metabolites M-1, M-7 and M-9) after IV SK-1404 | Predose to 96hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The peak plasma concentration (Cmax) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The time from dosing at which Cmax was apparent (Tmax) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The elapsed time from dosing at which the analyte was first quantifiable in a concentration vs time profile (Tlag) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The area under the concentration-time curve from dosing to the last measurable concentration (AUC(0-last)) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The area under the concentration-time curve from dosing extrapolated to infinity (AUC(0-inf)) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The percentage of AUC(0-inf) extrapolated beyond the last measured time point (AUC%extrap) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The terminal elimination rate constant calculated from the slope of the apparent elimination phase (lambda-z) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent terminal elimination half-life (T1/2) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The absolute bioavailability (F, PO vs IV from Part 1) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent total clearance (CL/F) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The apparent volume of distribution (Vd/F) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
The mean residence time (MRT) of SK-1404F and its active metabolites M-1, M-7 and M-9) after PO SK-1404 | Predose to 168hr
  Metabolite:parent ratios will be calculated for SK-1404F, M-1, M-7 and M-9
To collect further information about the safety and tolerability of IMP | Predose to 168hr
  By assessing physical examination, safety laboratory tests, vital signs, electrocardiograms (ECGs) and AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB BScMedSci, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No